CLINICAL TRIAL: NCT01694849
Title: A Multicentre, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GFT505 Once Daily on Steatohepatitis in Patients With Non-Alcoholic Steatohepatitis (NASH).
Brief Title: Phase IIb Study to Evaluate the Efficacy and Safety of GFT505 Versus Placebo in Patients With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Collaborators: Naturalpha (Industry); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-212-7; 2012-000295-42 (EudraCT Number)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: PPARs; NASH; Non-Alcoholic Steatohepatitis; Liver Diseases; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fibrosis | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GFT505 80mg (Experimental): Hard gelatin capsules dosed at 40mg, oral administration, 3 capsules per day before breakfast with a glass of water.
  Interventions: Drug: GFT505 80mg
- GFT505 120mg (Experimental): Hard gelatin capsules dosed at 40mg, oral administration, 3 capsules per day before breakfast with a glass of water.
  Interventions: Drug: GFT505 120mg
- Placebo (Placebo Comparator): hard gelatin capsules, oral administration, 3 capsules per day before breakfast with a glass of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFT505 80mg
  Arms: GFT505 80mg
Drug: GFT505 120mg
  Arms: GFT505 120mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Abdominal obesity and type-2 Diabetes are associated with chronic liver disorders resulting from the accumulation of fat in the liver (steatosis), which may progress towards hepatitis and possibly lead to cirrhosis and liver cancer. NAFLD (Non Alcoholic Fatty Liver Disease) is considered as the most common form of chronic liver disease in adults in the United States, Australia, Asia and Europe. In the USA, the estimated prevalence of NAFLD is 20-30% of the adult population.

Non-alcoholic Steatohepatitis (NASH) is a progressing form of NAFLD, which corresponds to hepatic steatosis associated with inflammation and liver cell injury upon microscopic examination of a liver biopsy. This condition may lead to advanced fibrosis and cirrhosis and deserves serious medical management. Up to now, there is no effective drug which has clearly demonstrated therapeutic efficacy which may help lifestyle and dietary recommendations in the resolution of NASH.

In this context, GENFIT is developing a new liver targeted drug candidate, GFT505, for the treatment of NASH and the reduction of multiple cardiometabolic risk factors associated with the metabolic syndrome and type 2 Diabetes.

This phase IIb study will evaluate the efficacy and safety of GFT505 80mg and 120mg once daily for 52 weeks on the reversal of NASH without worsening of fibrosis, based on liver biopsy assessments.

DETAILED DESCRIPTION:
The study duration per patient will be 80 weeks. A screening period (from 4 to 16 weeks) will precede a 52-week double-blind treatment period and a 3 months follow-up period.

The study will be conducted in 270 patients (90 patients in the placebo arm, 90 patients in the GFT505 80mg arm, and 90 patients in the GFT505 120mg arm).

Enrollment will be performed in two phases: during the first phase, the patients will receive either GFT505 at a dose of 80 mg either the placebo. An independent expert committee will review the safety data when 45 patients receiving the dose at 80 mg will have been treated for 6 months. The committee approval will be necessary to start the second phase, while the patients will receive either GFT505 at a dose of 80 mg, or GFT505 at a dose of 120 mg or the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (females must be either of non-child bearing potential or using an efficient double contraception). For male participants, contraceptive measures must be taken during the study, either by the male participant or his female partner.
* Body Mass Index ≤ 45 kg/m².
* Patients agree to have one liver biopsy during the screening period for diagnostic purpose (if no historical biopsy within 6 months before randomization is available) and one at the end of the treatment period for assessment of the treatment effects.
* For hypertensive patients, hypertension must be controlled by stable dose of anti-hypertensive medication for at least 2 months prior to screening (and the stable dose can be maintained throughout the study).
* Patients treated with vitamin E (>400IU/d), or Polyunsaturated fatty acids (>2g/day)or Ursodeoxycholic acid can be included if drugs are stopped at least 3 months prior to diagnostic liver biopsy and up to the end of the study.
* Histological confirmation of steatohepatitis on a diagnostic liver biopsy. Histological diagnostic is confirmed by central reading of the slides (steatosis > 5% + lobular inflammation, any grade + ballooning, any amount).
* For patients with Type 2 Diabetes, glycemia must be controlled (Glycosylated Haemoglobin A1c ≤8.5%). If glycemia is controlled by anti-diabetic drugs, qualitative change is not permitted within 6 months prior to randomization and should be avoided during the study. Treatments with metformin, Dipeptidyl Peptidase 4 inhibitors, Glucagon-like peptide-1 agonists, sulfamides, insulin are authorized. Sulfamides and insulin are permitted if glycemia is self-monitored by the patient.

Exclusion Criteria:

* Known heart failure (Grade I to IV of New York Heart Association classification).
* Weight loss of more than 5% within 6 months prior to randomization.
* History of bariatric surgery.
* Uncontrolled Blood Pressure.
* Type 1 diabetes patients.
* Patients who had an acute cardiovascular episode within the 6 months prior to screening, or with a history of coronary angioplasty, history of stroke, Transient Ischemic Attack, Coronary Heart Disease.
* Compensated and uncompensated cirrhosis. Notably, NASH patients with fibrosis stage = 4 according to the NASH CRN fibrosis staging system are excluded.
* Known alcohol and/or any other drug abuse or dependence in the last five years.
* Pregnant or lactating females.
* Other well documented causes of chronic liver disease
* Known intolerance or contra-indication to the list of excipients of GFT505.
* Evidence of any other unstable or, untreated clinically significant immunological, neoplastic, endocrine, haematological, gastrointestinal, neurological or psychiatric disorder.
* Positive HBsAg (Hepatitis B Surface Antigen), Positive anti-HIV, positive HCV-RNA (Hepatitis C Virus).
* Uncontrolled hypothyroidism defined as Thyroid Stimulating Hormone > 2X the upper limit of normal (ULN). Thyroid dysfunction controlled for at least 6 months prior to screening is permitted.
* Significant renal disease, including nephritic syndrome, chronic renal failure (defined as creatinine clearance < 60 mL/mn and serum creatinine >180 μmol/L).
* Unexplained serum creatine phosphokinase (CPK) > 3X the upper limit of normal (ULN). Patients with a reason for CPK elevation may have the measurement repeated prior to randomization; a CPK retest > 3X ULN leads to exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rémy HANF, PhD, Study Director — Development Director Genfit, France; Pr. Vlad RATZIU, M.D., Study Chair — International Coordinator - La Pitié-Salpêtrière Hospital - Paris 13, France; Pr. Arun SANYAL, M.D., Principal Investigator — National Coordinator -Virginia Commonwealth University - Richmond - USA; Dr. Sven FRANCQUE, M.D., Principal Investigator — National Coordinator - UZA - Edegem - Belgium; Dr. Jost PH DRENTH, MD, Ph.D, Principal Investigator — National Coordinator - UMC St Radboud Nijmegen - Nijmegen - The Netherlands; Pr. Michael Manns, M.D., Principal Investigator — National Coordinator - Medical School of Hannover - Hannover - Germany; Pr. Elisabetha BUGIANESI, M.D., Principal Investigator — National Coordinator - University of Torino - S. Giovanni Battista Hospital - Torino - Italy; Pr. Mihai VOICULESCU, M.D., Principal Investigator — National Coordinator - Center of Internal Medicine, Fundeni Clinical Institute - Bucharest - Romania; Pr. Manuel ROMERO-GOMEZ, M.D., Principal Investigator — National Coordinator - Valme University hospital - Sevilla - Spain; Pr. Quentin M. ANSTEE, M.D., Principal Investigator — National Coordinator - Freeman Hospital - Newcastle - UK
Locations (56):
- United States (19):
  - Site 920, Fresno, California
  - Site 903, La Jolla, California
  - Site 911, Aurora, Colorado
  - Site 912, Gainesville, Florida
  - Site 924, Atlanta, Georgia
  - Site 917, Atlanta, Georgia
  - Site 909, New Orleans, Louisiana
  - Site 921, Worcester, Massachusetts
  - Site 902, Detroit, Michigan
  - Site 927, New York, New York
  - Site 908, Durham, North Carolina
  - Site 919, Philadelphia, Pennsylvania
  - Site 916, Memphis, Tennessee
  - Site 913, Fort Sam Houston, Texas
  - Site 923, Houston, Texas
  - Site 906, San Antonio, Texas
  - Site 931, Salt Lake City, Utah
  - Site 930, Charlottesville, Virginia
  - Site 901, Richmond, Virginia
- Belgium (5):
  - Site 205, Brussels
  - Site 201, Edegem
  - Site 204, Ghent
  - Site 202, Haine-Saint-Paul
  - Site 203, Leuven
- France (12):
  - Site 106, Amiens
  - Site 102, Angers
  - Site 114, Clichy
  - Site 103, Lille
  - Site 113, Lyon
  - Site 111, Marseille
  - Site 108, Montpellier
  - Site 104, Nantes
  - Site 109, Nice
  - Site 112, Paris
  - Site 101, Paris
  - Site 107, Pessac
- Germany (2):
  - Site 405, Bonn
  - Site 404, Mainz
- Italy (4):
  - Site 507, Milan
  - Site 503, Palermo
  - Site 504, Roma
  - Site 501, Torino
- Netherlands (2):
  - Site 303, Amsterdam
  - Site 302, Nijmegen
- Romania (3):
  - Site 603, Bucharest
  - Site 601, Bucharest
  - Site 602, Bucharest
- Spain (5):
  - Site 703, Barcelona
  - Site 707, Majadahonda
  - Site 705, Málaga
  - Site 706, Santander
  - Site 701, Seville
- United Kingdom (4):
  - Site 802, Camberley
  - Site 808, Hull
  - Site 801, Newcastle upon Tyne
  - Site 803, Nottingham

REFERENCES:
- [Derived] Ratziu V, Harrison SA, Francque S, Bedossa P, Lehert P, Serfaty L, Romero-Gomez M, Boursier J, Abdelmalek M, Caldwell S, Drenth J, Anstee QM, Hum D, Hanf R, Roudot A, Megnien S, Staels B, Sanyal A; GOLDEN-505 Investigator Study Group. Elafibranor, an Agonist of the Peroxisome Proliferator-Activated Receptor-alpha and -delta, Induces Resolution of Nonalcoholic Steatohepatitis Without Fibrosis Worsening. Gastroenterology. 2016 May;150(5):1147-1159.e5. doi: 10.1053/j.gastro.2016.01.038. Epub 2016 Feb 11. PMID 26874076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the GFT505-212-7 study began in September 2012. This was a phase IIb, double-blind, randomized, placebo-controlled study conducted in three parallel groups: placebo, GFT505 80mg and GFT505 120mg (after DSMB review of 6 month safety data of the 80mg dose on at least 50% of participants) once daily for 52 weeks.
Pre-assignment Details: Random allocation was done in two phases. In the first study phase, participants were randomly allocated to GFT505 80 mg or placebo (ratio 2:1). In the second study phase (after Data and Safety Monitoring Board review of 6-month safety data of the 80-mg dose on at least 50% of participants), participants were assigned to GFT505 120 mg or placebo (ratio 2:1) in order to balance the 3 treatments in a 1:1:1 ratio basis.
Groups:
- GFT505 80mg: Hard gelatin capsules dosed at 40mg, oral administration.
  3 capsules per day (2 capsules of GFT505 40 mg and 1 capsule of placebo), before breakfast with a glass of water.
- GFT505 120mg: Hard gelatin capsules dosed at 40mg, oral administration.
  3 capsules of GFT505 40 mg per day, before breakfast with a glass of water.
- Placebo: Hard gelatin capsules, oral administration. Capsules of placebo were identical to capsules of investigational product to ensure double-blind conditions.
  3 placebo capsules per day, before breakfast with a glass of water.
Period: Treatment Period (Visit 2 to Visit 8)
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Started | 93 | 90 | 92
Randomized | 93 | 90 | 92
Randomised and Received Treatment (Full Analysis Set and Safety Set) | 93 | 89 | 92
Efficacy Evaluable Set (The Efficacy Evaluable Set included participants who completed the treatment period and did not have missing liver biopsies.) | 82 | 78 | 77
Completed | 84 | 79 | 78
Not Completed | 9 | 11 | 14
Not completed — Adverse Event | 6 | 7 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 1
Not completed — Randomized and not treated | 0 | 1 | 0
Period: Follow-up Period (to Visit 9)
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Started | 84 | 79 | 78
Completed | 83 | 76 | 77
Not Completed | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo | Total
Number analyzed (Participants) | 93 | 89 | 92 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] — Data collected at Visit 1
  years | 53.26 (11.02) | 52.88 (11.63) | 52.88 (11.99) | 53.01 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Data collected at Visit 1
  Participants
    Female | 44 | 42 | 37 | 123
    Male | 49 | 47 | 55 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data collected at Visit 1
  Participants
    Race: Caucasian | 88 | 71 | 85 | 244
    Race: Black | 2 | 5 | 3 | 10
    Race: Asian | 0 | 6 | 1 | 7
    Race: Other | 3 | 7 | 3 | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Data collected at Visit 2
  kg/m^2 | 31.80 (5.20) | 31.04 (4.39) | 30.91 (4.15) | 31.25 (4.61)
Type 2 diabetes [Number; unit: participants]
  Type 2 diabetes (Yes) | 37 | 37 | 33 | 107
  Type 2 diabetes (No) | 56 | 52 | 59 | 167
Height [Mean (Standard Deviation); unit: cm] — Data collected at Visit 1
  cm | 167.77 (9.30) | 170.21 (10.69) | 169.21 (10.23) | 169.05 (10.09)
Weight [Mean (Standard Deviation); unit: kg] — Data collected at Visit 2
  kg | 89.62 (17.76) | 90.15 (15.57) | 88.72 (15.79) | 89.49 (16.36)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Data collected at Visit 2
  cm | 106.41 (13.09) | 106.26 (10.28) | 104.68 (10.52) | 105.78 (11.37)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With Disappearance of Steatohepatitis Without Worsening of Fibrosis (ie, Participants no Longer Meeting the Criteria for Steatohepatitis)
Description: Percentage of responders from baseline to Week 52 defined by the disappearance of steatohepatitis (ie, participants no longer meeting the criteria for steatohepatitis) without worsening of fibrosis.
  Worsening of fibrosis was evaluated using Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) fibrosis staging system and defined as:
  * Progression to stage 3 or 4 for participants at stage 0, 1 or 2 on diagnostic liver biopsy
  * Progression to stage 4 for participants at stage 3 on diagnostic liver biopsy
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Analysis was done of the efficacy evaluable sample, (Efficacy Evaluable Set) formed by participants with liver biopsy available at end-of-treatment and considered as the Intent to Treat population in the protocol. Robustness analysis was also performed in the Full Analysis Set, formed by all randomized participants that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 89 | 92
Participants
  Efficacy evaluable set: number analyzed (Participants) | 82 | 78 | 77
  Efficacy evaluable set: Responders | 21 | 19 | 16
  Efficacy evaluable set: Non-responders | 61 | 59 | 61
  Full analysis set: Responders | 21 | 19 | 16
  Full analysis set: Non-responders | 72 | 70 | 76
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; H_01: OR_80 less than or equal to 1 versus H_11 : OR_80 greater than 1 H_02: OR_120 less than or equal to 1 versus H_12 : OR_120 greater than 1; Test type: Superiority; p = 0.8539, Regression, Logistic — To deal with multiplicity of comparisons, a step-down approach was adopted to control the type I error to 0.05. The contrast GFT120 mg versus placebo was examined first. If not significant the GFT 80mg versus placebo contrast was not examined; Baseline NAS, Log transformed baseline aspartate aminotransferase and baseline plasminogen activator inhibitor 1 values; Odds Ratio (OR) = 1.092, 95% CI 2-sided [0.427 to 2.795] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8160, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Baseline NAS, Log transformed baseline aspartate aminotransferase and baseline plasminogen activator inhibitor 1 values; Odds Ratio (OR) = 0.897, 95% CI 2-sided [0.361 to 2.232] — Standard error of the estimate

2. Secondary Outcome: Change From Baseline to Week 52 in Non-alcoholic Fatty Liver Disease Activity Score
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg the change from baseline to Week 52, in Non-alcoholic Fatty Liver Disease Activity Score (NAS score).
  NAS score is a composite score equal to the sum of the steatosis grade (0 to 3), lobular inflammation grade (0 to 3) and hepatocellular ballooning grade (0 to 2). The overall scale of the NAS is 0 to 8, with higher scores indicating more severe disease. The outcome measure, change from baseline in NAFLD Activity Score (NAS), has a possible range from -8 to +8, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: NAS score
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
NAS score | -0.65 (1.33) | -0.64 (1.68) | -0.45 (1.34)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; H0: difference in least squares (LS) mean change from baseline equal to 0 H1: difference in LS mean change from baseline not equal to 0 Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.225, Mixed Models Analysis; Baseline Non-Alcoholic Fatty Liver Disease Activity Score; difference in least square mean change = -0.27, 95% CI 2-sided [-0.75 to 0.2] — Standard error of the least squares mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.254, Mixed Models Analysis; Baseline Non-Alcoholic Fatty Liver Disease Activity Score; Difference in least square mean change = -0.28, 95% CI 2-sided [-0.76 to 0.2] — Standard error of the least squares mean

3. Secondary Outcome: Number of Participants With Change From Baseline to Week 52 in Non-alcoholic Fatty Liver Disease Activity Score of at Least 2 Points
Description: To evaluate the number of participants with at least a 2 point decrease from baseline in Non-alcoholic Fatty Liver Disease Activity Score (NAS) after 52 weeks of daily administration of GFT505 80mg or 120mg. The NAS refers to the severity of ongoing liver injury as assessed by a liver biopsy and is used to assess the activity of the disease. It is based on the NASH CRN methodology for scoring the severity of steatosis (score of 0 to 3), inflammation (score of 0 to 3), and hepatocellular ballooning (score of 0 to 2), with a maximum score of 8. A total NAS score of five or greater correlates with the diagnosis of steatohepatitis.
  In table below for raw "Mild (Nonalcoholic Fatty Liver Disease Activity Score 3)" and the column "GFT505 80mg" the result should be read as : 2 participants (out of 10 participants analysed with a baseline NAS at 3) had at Least 2 points decrease on their NAS after 52 weeks of daily administration of GFT505 80mg. It corresponds to 20% (2 out of 10).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Count of Participants; unit: Participants
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Participants
  Mild (Non-alcoholic Fatty Liver Disease Activity Score 3): number analyzed (Participants) | 10 | 11 | 14
  Mild (Non-alcoholic Fatty Liver Disease Activity Score 3) | 2 | 2 | 5
  Moderate (Non-alcoholic Fatty Liver Disease Activity Score 4-5): number analyzed (Participants) | 49 | 40 | 41
  Moderate (Non-alcoholic Fatty Liver Disease Activity Score 4-5) | 11 | 12 | 9
  Severe (Non-alcoholic Fatty Liver Disease Activity Score 6-8): number analyzed (Participants) | 23 | 27 | 22
  Severe (Non-alcoholic Fatty Liver Disease Activity Score 6-8) | 8 | 12 | 7
  Total | 21 | 26 | 21
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.8586, Regression, Logistic; Baseline Non-Alcoholic Fatty Liver Disease Activity Score; Odds Ratio (OR) = 1.073, 95% CI 2-sided [0.493 to 2.339] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.2265, Regression, Logistic; Baseline Non-Alcoholic Fatty Liver Disease Activity Score; Odds Ratio (OR) = 1.601, 95% CI 2-sided [0.747 to 3.432] — Standard error of the estimate

4. Secondary Outcome: Number of Participants With Decrease in Steatosis Score of at Least 1 Point Between Baseline and Week 52
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, number of participants with a decrease in steatosis score of at least 1 point between baseline and Week 52.
  Steatosis is assessed by a liver biopsy and evaluated on a scale of 0 to 3 with higher scores indicating more severe steatosis. A score of 0 indicating a lower severity with low parenchymal involvement (<5%), while a score of 3 is indicative of higher involvment/severity (> 66%).
  In below table and for helping how results are reported, as an example for raw "Mild (Nonalcoholic Fatty Liver Disease Activity Score 3)" and the column "GFT505 80mg" the result should be read as : 1 participants (out of 10 participants analysed with a baseline NAS at 3) had at least 1 point decrease Steatosis Score after 52 weeks of daily administration of GFT505 80mg. It corresponds to 10% (1 out of 10).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Count of Participants; unit: Participants
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Participants
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3): number analyzed (Participants) | 10 | 11 | 14
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3) | 1 | 1 | 0
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5): number analyzed (Participants) | 49 | 40 | 41
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5) | 13 | 10 | 12
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8): number analyzed (Participants) | 23 | 27 | 22
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8) | 3 | 10 | 3
  Total | 17 | 21 | 15
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.5231, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 0.723, 95% CI 2-sided [0.267 to 1.958] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.8459, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 1.102, 95% CI 2-sided [0.415 to 2.924] — Standard error of the estimate

5. Secondary Outcome: Number of Participants With Decrease in Lobular Inflammation Score of at Least 1 Point Between Baseline and Week 52
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, number of participants with a decrease in lobular inflammation score of at least 1 point between baseline and Week 52.
  Lobular inflammation is assessed by a liver biopsy and evaluated on a scale of 0 to 3. A score of 0 indicating the absence of inflammation loci, while a score of 3 is indicative of a higher degree of inflammation with more than 4 inflammation loci 200 x field.
  In below table and for helping how results are reported, as an example for raw "Mild (Nonalcoholic Fatty Liver Disease Activity Score 3)" and the column "GFT505 80mg" the result should be read as : 1 participants (out of 10 participants analysed with a baseline NAS at 3) had at least 1 point decrease of Lobular Inflammation Score after 52 weeks of daily administration of GFT505 80mg. It corresponds to 10% (1 out of 10).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Count of Participants; unit: Participants
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Participants
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3): number analyzed (Participants) | 10 | 11 | 14
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3) | 1 | 2 | 7
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5): number analyzed (Participants) | 49 | 40 | 41
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5) | 10 | 11 | 8
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8): number analyzed (Participants) | 23 | 27 | 22
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8) | 14 | 16 | 12
  Total | 25 | 29 | 27
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.5229, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 0.638, 95% CI 2-sided [0.161 to 2.529] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.5646, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 1.433, 95% CI 2-sided [.421 to 4.875] — Standard error of the estimate

6. Secondary Outcome: Title: Number of Participants With Decrease in Ballooning Score of at Least 1 Point Between Baseline and Week 52
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, number of participants with a decrease in ballooning score of at least 1 point between baseline and Week 52.
  Ballooning is assessed by a liver biopsy and evaluated on a scale of 0 to 2 with higher scores indicating more severe ballooning (0: No ballooned cells, 1: Few [rare but definite] ballooned hepatocytes; 2: Many ballooned cells/prominent ballooning).
  In below table and for helping how results are reported, as an example for raw "Mild (Nonalcoholic Fatty Liver Disease Activity Score 3)" and the column "GFT505 80mg" the result should be read as : 4 participants (out of 10 participants analysed with a baseline NAS at 3) had at least 1 point decrease of Ballooning Score after 52 weeks of daily administration of GFT505 80mg. It corresponds to 10% (1 out of 10).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Count of Participants; unit: Participants
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Participants
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3): number analyzed (Participants) | 10 | 11 | 14
  Mild (Non-Alcoholic Fatty Liver Disease Activity Score 3) | 4 | 3 | 6
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5): number analyzed (Participants) | 49 | 40 | 41
  Moderate (Non-Alcoholic Fatty Liver Disease Activity Score 4-5) | 17 | 15 | 13
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8): number analyzed (Participants) | 23 | 27 | 22
  Severe (Non-Alcoholic Fatty Liver Disease Activity Score 6-8) | 10 | 12 | 5
  Total | 31 | 30 | 24
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.1983, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 0.382, 95% CI 2-sided [0.088 to 1.656] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 1.0000, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.288 to 3.466] — Standard error of the estimate

7. Secondary Outcome: Changes From Baseline to Week 52 in the Stages of Fibrosis
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in stages of fibrosis (based on Non-Alcoholic Steatohepatitis Clinical Research Network [NASH CRN] scoring).
  Fibrosis is assessed on a scale of 0 to 4 with higher scores indicating more severe fibrosis.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: Change in fibrosis score
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Change in fibrosis score | -0.23 (0.84) | -0.06 (0.96) | -0.23 (0.90)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.3543, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 0.653, 95% CI 2-sided [0.265 to 1.609] — Standard error of the estimate
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Population with baseline Non-Alcoholic Fatty Liver Disease Activity Score greater than or equal to 4; Test type: Superiority; p = 0.5780, Regression, Logistic; Baseline value of the analyzed parameter; Odds Ratio (OR) = 1.270, 95% CI 2-sided [0.547 to 2.953] — Standard error of the estimate

8. Secondary Outcome: Changes From Baseline to Visit 8 (Week 52) in Liver Enzymes
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to week 52, in liver enzymes.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
U/L
  Gamma-glutamyl transferase | -24.32 (36.39) | -20.59 (40.45) | 6.22 (50.64)
  Aspartate transaminase | 1.88 (27.76) | -1.37 (24.74) | -1.32 (16.63)
  Alanine aminotransferase | -7.02 (36.21) | -12.54 (44.72) | -3.26 (24.67)
  Alkaline phosphatases | -18.82 (13.23) | -20.44 (16.47) | 3.44 (13.16)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Change in aspartate transaminase (U/L); Test type: Superiority; p = 0.711, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 1.24, 95% CI 2-sided [-5.33 to 7.81] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Change in aspartate transaminase (U/L); Test type: Superiority; p = 0.78, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.94, 95% CI 2-sided [-7.58 to 5.7] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Change in alanine aminotransferase (U/L); Test type: Superiority; p = 0.221, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -6.13, 95% CI 2-sided [-15.97 to 3.71] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Change in alanine aminotransferase (U/L); Test type: Superiority; p = 0.062, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -9.45, 95% CI 2-sided [-19.4 to 0.49] — Standard error of the least square mean
Statistical Analysis 5: Comparison: GFT505 80mg vs Placebo; Change in Alkaline phosphatases (U/L); Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -23.02, 95% CI 2-sided [-27.16 to -18.88] — Standard error of the least square mean
Statistical Analysis 6: Comparison: GFT505 120mg vs Placebo; Change in Alkaline phosphatases (U/L); Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -23.85, 95% CI 2-sided [-28.04 to 2.12] — Standard error of the least square mean
Statistical Analysis 7: Comparison: GFT505 80mg vs Placebo; Change in Gamma-glutamyl transferase (U/L); Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -31.41, 95% CI 2-sided [-43.78 to -19.05] — Standard error of the least square mean
Statistical Analysis 8: Comparison: GFT505 120mg vs Placebo; Change in Gamma-glutamyl transferase (U/L); Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -29.31, 95% CI 2-sided [-41.84 to -16.77] — Standard error of the least square mean

9. Secondary Outcome: Changes From Baseline to Visit 8 (Week 52) in Aspartate Transaminase/Alanine Aminotransferase Ratio
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to week 52, in aspartate transaminase/alanine aminotransferase ratio
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
ratio | 0.15 (0.21) | 0.20 (0.25) | 0.01 (0.25)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.14, 95% CI 2-sided [0.06 to 0.21] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.19, 95% CI 2-sided [0.11 to 0.26] — Standard error of the least square mean

10. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: CK 18-M65
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in CK 18-M65 (non-invasive markers of fibrosis and steatosis).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
U/L | 104.4 (804.96) | -185.01 (658.14) | -45.53 (437.21)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.095, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 141.78, 95% CI 2-sided [-24.99 to 308.55] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.412, Mixed Models Analysis — Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -70.57, 95% CI 2-sided [-239.85 to 98.71] — Standard error of the least square mean

11. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: CK18 M30
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in CK18 M30 (non-invasive markers of fibrosis and steatosis).
  Participants with missing data for CK18 M30 at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 76
pmol/L | -28.08 (574.50) | -66.40 (432.02) | -51.39 (349.64)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.592, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 32.39, 95% CI 2-sided [-86.63 to 151.42] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.61, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 31.35, 95% CI 2-sided [-89.42 to 152.12] — Standard error of the least square mean

12. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Adiponectin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in adiponectin (non-invasive markers of fibrosis and steatosis).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
μg/mL | 4.98 (20.25) | 1.90 (8.34) | 2.54 (9.48)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.459, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 1.67, 95% CI 2-sided [-2.77 to 6.11] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.764, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.67, 95% CI 2-sided [-5.06 to 3.72] — Standard error of the least square mean

13. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Ferritin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in ferritin (non-invasive markers of fibrosis and steatosis).
  Participants with missing data for Ferritin at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 77 | 76
μg/L | -23.52 (145.61) | -19.68 (81.91) | -19.26 (122.57)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.466, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -12.92, 95% CI 2-sided [-47.79 to 21.95] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.745, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -5.82, 95% CI 2-sided [-41.07 to 29.42] — Standard error of the least square mean

14. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: FG19 and FG21
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in FG19 and FG21 (non-invasive markers of fibrosis and steatosis).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
pg/mL
  FG19 | -27.25 (94.19) | -26.03 (91.59) | 11.64 (87.10)
  FG21 | 258.74 (1138.36) | 319.68 (433.63) | 73.05 (360.41)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; FG19; Test type: Superiority; p = 0.018, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -26.57, 95% CI 2-sided [-48.59 to -4.54] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; FG19; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -40.39, 95% CI 2-sided [-62.61 to -18.17] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; FG21; Test type: Superiority; p = 0.101, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 190.07, 95% CI 2-sided [-37.38 to 417.52] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; FG21; Test type: Superiority; p = 0.052, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 228.33, 95% CI 2-sided [-2.16 to 458.82] — Standard error of the least square mean

15. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Alpha2 Macroglobulin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in alpha2 macroglobulin (a non-invasive marker of fibrosis and steatosis).
  Participants with missing data for Alpha2 Macroglobulin at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 77 | 76
g/L | -0.14 (0.29) | -0.26 (0.36) | 0.01 (0.28)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.14, 95% CI 2-sided [-0.29 to -0.01] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.24, 95% CI 2-sided [-0.34 to -0.15] — Standard error of the least square mean

16. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Hyaluronic Acid, N-terminal Pro-peptide of Collagen Type III (PIIINP), and Tissue Inhibitor of Matrix Metalloprotease-1 (TIMP-1)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in hyaluronic acid, N-terminal pro-peptide of collagen type III (PIIINP), and tissue inhibitor of matrix metalloprotease-1 (TIMP-1) (non-invasive markers of fibrosis and steatosis).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
ng/mL
  Hyaluronic acid: number analyzed (Participants) | 82 | 78 | 76
  Hyaluronic acid | 26.12 (230.97) | 12.14 (48.04) | 12.49 (48.68)
  PIIINP: number analyzed (Participants) | 81 | 78 | 77
  PIIINP | -0.50 (3.43) | -0.57 (3.75) | 0.29 (4.87)
  TIMP-1: number analyzed (Participants) | 81 | 78 | 77
  TIMP-1 | 15.21 (35.38) | -6.32 (39.75) | 9.08 (49.54)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Hyaluronic acid; Test type: Superiority; p = 0.203, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -16.54, 95% CI 2-sided [-42.07 to 8.98] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.603, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -6.79, 95% CI 2-sided [-32.49 to 18.9] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; PIIINP; Test type: Superiority; p = 0.235, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.73, 95% CI 2-sided [-1.95 to 0.48] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; PIIINP; Test type: Superiority; p = 0.193, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.81, 95% CI 2-sided [-2.04 to 0.41] — Standard error of the least square mean
Statistical Analysis 5: Comparison: GFT505 80mg vs Placebo; TIMP-1; Test type: Superiority; p = 0.348, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 6.21, 95% CI 2-sided [-6.81 to 19.22] — Standard error of the least square mean
Statistical Analysis 6: Comparison: GFT505 120mg vs Placebo; TIMP-1; Test type: Superiority; p = 0.029, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -14.66, 95% CI 2-sided [-27.81 to 1.51] — Standard error of the least square mean

17. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Fibrotest
Description: Fibrotest combines α2-macroglobulin (a2m), apolipoprotein A1 (aA1), total bilirubin (BIL), haptoglobin (h), GGT, and ALT with adjustment for age and gender. Fibrotest is calculated as: z = 4.467 x log(a2m) - 1.357 x log(h) + 1.017 x log(GGT) + 0.0281 x Age + 1.737 x log(BIL) - 1.184 x (aA1) + 0.301 x Gender - 5.54 where Gender = 1 for male and Gender = 0 for female. The score is then: 1/(1+e^-z). Calculated score range from 0 (no fibrosis) to 1 (severe fibrosis or cirrhosis) In below table for "Fibrotest" and for column "GFT505 80mg" the result should be read as: the mean of change from baseline to week 52 of Fibrotest calculated in 81 participants is -0.06 with a standard deviation of 0.08.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
score on a scale | -0.06 (0.08) | -0.07 (0.09) | -0.01 (0.10)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.05, 95% CI 2-sided [-0.07 to -0.02] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.05, 95% CI 2-sided [-0.08 to -0.02] — Standard error of the least square mean

18. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Steatotest
Description: SteatoTest combines α2-macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, GGT, fasting glucose, triglycerides, cholesterol, and ALT, adjusted for patient's age, sex, weight, and height. Patented formula. Calculated score range from 0 (no steatosis) to 1 (severe steatosis) In below table for "Steatotest" and for column "GFT505 80mg" the result should be read as: the mean of change from baseline to week 52 of Steatotest calculated in 81 participants is -0.09 with a standard deviation of 0.11.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 77 | 74
score on a scale | -0.09 (0.11) | -0.08 (0.15) | 0.03 (0.11)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.11, 95% CI 2-sided [-0.15 to -0.07] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.11, 95% CI 2-sided [-0.15 to -0.07] — Standard error of the least square mean

19. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Angulo Index or Non-Alcoholic Fatty Liver Disease Fibrosis Score
Description: Angulo Index or Non-Alcoholic Fatty Liver Disease Fibrosis Score is based on age, hyperglycemia, BMI, platelet count, albumin level, and AST/ALT ratio. Score is calculated using the following formula: -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m^2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet (×10^9/l) - 0.66 × albumin (g/dl). A score of <-1.455 indicates no advanced fibrosis and a score of >0.676 indicates liver fibrosis.
  In below table for "Angulo index" and for column "GFT505 80mg" the result should be read as: the mean of change from baseline to week 52 of Angulo index calculated in 82 participants is 0.06 with a standard deviation of 0.53.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 75 | 76
score on a scale | 0.06 (0.53) | -0.26 (0.57) | -0.01 (0.51)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.471, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.06, 95% CI 2-sided [-0.11 to 0.23] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.25, 95% CI 2-sided [-0.42 to -0.08] — Standard error of the least square mean

20. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Enhanced Liver Fibrosis (ELF)
Description: Enhanced Liver Fibrosis (ELF) combines measurements of tissue inhibitor of metalloprotein-ases-1 (TIMP-1), amino-terminal propeptide of type III procollagen (PIIINP), and hyaluronic acid (HA) . The ELF score is calculated as : 2.278 + 0.851 ln (HA) + 0.751 ln (PIIINP) + 0.394 ln (TIMP-1). ELF score range from An ELF score of less than 7.7 indicates no fibrosis. An ELF score greater than or equal to 9.8 indicates severe fibrosis. An ELF score of 11.3 or greater indicates cirrhosis. A decrease in ELF score represents a positive outcome In below table for "Enhanced Liver Fibrosis" and for column "GFT505 80mg" the result should be read as : the mean of change from baseline to week 52 of Enhanced Liver Fibrosis calculated in 81 analysed participants is -0.01 with a standard deviation of 0.54.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 78 | 76
score on a scale | -0.01 (0.54) | -0.01 (0.64) | 0.08 (0.70)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.457, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.07, 95% CI 2-sided [-0.27 to 0.12] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.428, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean = -0.08, 95% CI 2-sided [-0.28 to 0.12] — Standard error of the least square mean

21. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Fatty Liver Index (FLI)
Description: The Fatty Liver Index (FLI) combines triglycerides, BMI, GGT and Waist circumference. FLI is calculated as : (e0.953×loge[triglycerides]+0.139× Body Mass Index[BMI]+0.718×loge Gamma- Glutamyl Transferase [GGT]+0.053×waistcircumference-15.745)/ (1 +e0.953×loge[triglycerides]+0.139×BMI+0.718×loge [GGT]+0.053×waistcircumference-15.745) × 100. Calculated index range from 0 to 100. FLI score below 30 indicate absence of Fatty Liver and FLI Score of 60 and above indicates presence of Fatty Liver.
  In below table for "Fatty Liver Index" and for column "GFT505 80mg" the result should be read as : the mean of change from baseline to week 52 of Fatty Liver Index calculated in 82 analysed participants is -7.94 with a standard deviation of 11.74.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 77 | 76
score on a scale | -7.94 (11.74) | -7.81 (14.29) | 1.34 (11.65)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -9.22, 95% CI 2-sided [-13.19 to -5.24] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -9.08, 95% CI 2-sided [-13.12 to -5.04] — Standard error of the least square mean

22. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Fibrometer
Description: Fibrometer combines Platelets, AST, ALT, ferritin, glucose (fasting plasma), Weight and gender. Patented formula. Score ranges from 0 (no fibrosis) to 1 (severe fibrosis or cirrhosis) In below table for "Fibrometer" and for column "GFT505 80mg" the result should be read as : the mean of change from baseline to week 52 of Fibrometer calculated in 81 analysed participants is 0.04 with a standard deviation of 0.23.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 74 | 71
score on a scale | 0.04 (0.23) | 0 (0.20) | 0.02 (0.22)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.531, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.02, 95% CI 2-sided [-0.05 to 0.09] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.638, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.02, 95% CI 2-sided [-0.08 to 0.05] — Standard error of the least square mean

23. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Total Bilirubin and Conjugated Bilirubin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in total bilirubin and conjugated bilirubin (non-invasive markers of fibrosis and steatosis).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
umol/L
  Total bilirubin | -1.53 (3.66) | -1.38 (4.85) | -1.46 (3.77)
  Conjugated bilirubin | -0.35 (1.26) | -0.15 (1.24) | -0.26 (1.05)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Total bilirubin; Test type: Superiority; p = 0.831, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.14, 95% CI 2-sided [-1.39 to 1.12] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Total bilirubin; Test type: Superiority; p = 0.754, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.2, 95% CI 2-sided [-1.07 to 1.47] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Conjugated Bilirubin; Test type: Superiority; p = 0.848, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.03, 95% CI 2-sided [-0.36 to 0.3] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Conjugated Bilirubin; Test type: Superiority; p = 0.511, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.11, 95% CI 2-sided [-0.22 to 0.45] — Standard error of the least square mean

24. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: Prothrombin Ratio
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in prothrombin ratio (non-invasive marker of fibrosis and steatosis).
  The Prothrombin ratio is the ratio of a participants measured prothrombin time (in seconds) to the normal laboratory reference prothrombin time.
  Participants with missing data for Prothrombin ratio at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 76 | 75
ratio | -3.85 (11.57) | 1.29 (10.03) | 0.51 (14.28)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.075, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -2.83, 95% CI 2-sided [-5.95 to 0.29] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.491, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.11, 95% CI 2-sided [-4.29 to 2.07] — Standard error of the least square mean

25. Secondary Outcome: Changes From Baseline to Week 52 in Non-invasive Markers of Fibrosis and Steatosis: International Normalized Ratio (INR)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg, the changes from baseline to week 52, in international normalized ratio (INR; non-invasive marker of fibrosis and steatosis).
  Participants with missing data for International Normalized Ratio (INR) at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 76 | 75
ratio | 0.03 (0.09) | -0.01 (0.08) | 0.03 (0.39)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.393, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.03, 95% CI 2-sided [-0.1 to 0.04] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.289, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.04, 95% CI 2-sided [-0.11 to 0.03] — Standard error of the least square mean

26. Secondary Outcome: Changes From Baseline to Week 52 in Lipid Parameters (Cardiovascular Risk Profile)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to week 52, in lipid parameters (used to assess cardiovascular risk)
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
mmol/L
  Triglycerides | -0.33 (0.76) | -0.48 (0.90) | 0.16 (1.12)
  Cholesterol | -0.42 (0.78) | -0.42 (0.72) | 0.02 (0.66)
  Non-high Density Lipoproteins Cholesterol | -0.45 (0.79) | -0.47 (0.71) | 0.07 (0.67)
  High Density Lipoproteins Cholesterol | 0.02 (0.17) | 0.06 (0.23) | -0.06 (0.21)
  Very Low Density Lipoproteins Cholesterol: number analyzed (Participants) | 82 | 75 | 74
  Very Low Density Lipoproteins Cholesterol | -0.17 (0.28) | -0.17 (0.32) | 0.05 (0.23)
  Low Density Lipoproteins Cholesterol: number analyzed (Participants) | 82 | 75 | 74
  Low Density Lipoproteins Cholesterol | -0.27 (0.70) | -0.25 (0.61) | -0.01 (0.51)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Triglycerides; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.47, 95% CI 2-sided [-0.73 to -0.21] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Triglycerides; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.55, 95% CI 2-sided [-0.81 to -0.29] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Cholesterol; Test type: Superiority; p = 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.35, 95% CI 2-sided [-0.56 to -0.14] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.43, 95% CI 2-sided [-0.64 to -0.23] — Standard error of the least square mean
Statistical Analysis 5: Comparison: GFT505 80mg vs Placebo; Non-high Density Lipoproteins Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.46, 95% CI 2-sided [-0.67 to -0.24] — Standard error of the least square mean
Statistical Analysis 6: Comparison: GFT505 120mg vs Placebo; Non-high Density Lipoproteins Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.54, 95% CI 2-sided [-0.75 to -0.32] — Standard error of the least square mean
Statistical Analysis 7: Comparison: GFT505 80mg vs Placebo; High Density Lipoproteins Cholesterol; Test type: Superiority; p = 0.005, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.09, 95% CI 2-sided [0.03 to 0.15] — Standard error of the least square mean
Statistical Analysis 8: Comparison: GFT505 120mg vs Placebo; High Density Lipoproteins Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.11, 95% CI 2-sided [0.05 to 0.17] — Standard error of the least square mean
Statistical Analysis 9: Comparison: GFT505 80mg vs Placebo; Very Low Density Lipoproteins Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.18, 95% CI 2-sided [-0.26 to -0.11] — Standard error of the least square mean
Statistical Analysis 10: Comparison: GFT505 120mg vs Placebo; Very Low Density Lipoproteins Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.17, 95% CI 2-sided [-0.25 to -0.09] — Standard error of the least square mean
Statistical Analysis 11: Comparison: GFT505 80mg vs Placebo; Low Density Lipoproteins Cholesterol; Test type: Superiority; p = 0.031, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.2, 95% CI 2-sided [-0.38 to -0.02] — Standard error of the least square mean
Statistical Analysis 12: Comparison: GFT505 120mg vs Placebo; Low Density Lipoproteins Cholesterol; Test type: Superiority; p = 0.009, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.24, 95% CI 2-sided [-0.42 to -0.06] — Standard error of the least square mean

27. Secondary Outcome: Changes From Baseline to Week 52 in Outcomes Related to Biochemistry
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to week 52, in secondary outcomes related to biochemistry
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
mg/dL
  Apo A1 | 1.63 (15.59) | 2.85 (20.42) | -3.90 (16.53)
  Apo B | -12.80 (20.87) | -8.42 (16.03) | 0.94 (14.29)
  Apo AII: number analyzed (Participants) | 66 | 65 | 60
  Apo AII | -0.15 (6.63) | 4.25 (4.36) | -3.36 (4.82)
  Apo CIII: number analyzed (Participants) | 66 | 65 | 60
  Apo CIII | -1.79 (3.91) | -0.69 (3.42) | 0.77 (4.30)
  Apo CIII/B: number analyzed (Participants) | 66 | 65 | 60
  Apo CIII/B | -1.44 (2.98) | -0.65 (2.98) | 0.53 (3.05)
  Apo CIII/nonB: number analyzed (Participants) | 66 | 65 | 60
  Apo CIII/nonB | -0.35 (1.79) | -0.04 (0.76) | 0.24 (2.53)
  Small dense Low Density Lipoproteins: number analyzed (Participants) | 71 | 69 | 69
  Small dense Low Density Lipoproteins | -2.09 (11.02) | -2.62 (6.08) | 0.60 (7.52)
  Lp(a): number analyzed (Participants) | 66 | 65 | 60
  Lp(a) | -0.57 (12.24) | -0.91 (13.75) | 0.80 (4.46)
  Apo E: number analyzed (Participants) | 66 | 65 | 60
  Apo E | -1.72 (2.75) | -1.38 (2.99) | -0.29 (3.67)
  Apo E/B: number analyzed (Participants) | 66 | 65 | 60
  Apo E/B | -1.43 (2.43) | -1.48 (2.64) | -0.21 (2.59)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Apo A1; Test type: Superiority; p = 0.038, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 5.73, 95% CI 2-sided [0.31 to 11.14] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Apo A1; Test type: Superiority; p = 0.012, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 7.07, 95% CI 2-sided [1.59 to 12.55] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Apo B; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -12.41, 95% CI 2-sided [-17.56 to -7.25] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Apo B; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -9.61, 95% CI 2-sided [-14.81 to -4.41] — Standard error of the least square mean
Statistical Analysis 5: Comparison: GFT505 80mg vs Placebo; Apo AII; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 3.55, 95% CI 2-sided [2.14 to 4.96] — Standard error of the least square mean
Statistical Analysis 6: Comparison: GFT505 120mg vs Placebo; Apo AII; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 6.1, 95% CI 2-sided [4.67 to 7.53] — Standard error of the least square mean
Statistical Analysis 7: Comparison: GFT505 80mg vs Placebo; Apo CIII; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -2.27, 95% CI 2-sided [-3.29 to -1.25] — Standard error of the least square mean
Statistical Analysis 8: Comparison: GFT505 120mg vs Placebo; Apo CIII; Test type: Superiority; p = 0.004, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.5, 95% CI 2-sided [-2.52 to -0.49] — Standard error of the least square mean
Statistical Analysis 9: Comparison: GFT505 80mg vs Placebo; Apo CIII/B; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.78, 95% CI 2-sided [-2.63 to -0.92] — Standard error of the least square mean
Statistical Analysis 10: Comparison: GFT505 120mg vs Placebo; Apo CIII/B; Test type: Superiority; p = 0.009, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.15, 95% CI 2-sided [-2 to -0.29] — Standard error of the least square mean
Statistical Analysis 11: Comparison: GFT505 80mg vs Placebo; Apo CIII/nonB; Test type: Superiority; p = 0.002, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.46, 95% CI 2-sided [-0.75 to -0.17] — Standard error of the least square mean
Statistical Analysis 12: Comparison: GFT505 120mg vs Placebo; Apo CIII/nonB; Test type: Superiority; p = 0.008, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.39, 95% CI 2-sided [-0.68 to -0.1] — Standard error of the least square mean
Statistical Analysis 13: Comparison: GFT505 80mg vs Placebo; Small dense Low Density Lipoproteins; Test type: Superiority; p = 0.069, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -2.35, 95% CI 2-sided [-4.89 to 0.19] — Standard error of the least square mean
Statistical Analysis 14: Comparison: GFT505 120mg vs Placebo; Small dense Low Density Lipoproteins; Test type: Superiority; p = 0.01, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -3.39, 95% CI 2-sided [-5.95 to -0.84] — Standard error of the least square mean
Statistical Analysis 15: Comparison: GFT505 80mg vs Placebo; Lp(a); Test type: Superiority; p = 0.549, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.84, 95% CI 2-sided [-1.93 to 3.61] — Standard error of the least square mean
Statistical Analysis 16: Comparison: GFT505 120mg vs Placebo; Lp(a); Test type: Superiority; p = 0.728, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.49, 95% CI 2-sided [-2.28 to 3.26] — Standard error of the least square mean
Statistical Analysis 17: Comparison: GFT505 80mg vs Placebo; Apo E; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.38, 95% CI 2-sided [-2.14 to -0.61] — Standard error of the least square mean
Statistical Analysis 18: Comparison: GFT505 120mg vs Placebo; Apo E; Test type: Superiority; p = 0.004, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.12, 95% CI 2-sided [-1.89 to -0.36] — Standard error of the least square mean
Statistical Analysis 19: Comparison: GFT505 80mg vs Placebo; Apo E/B; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.18, 95% CI 2-sided [-1.82 to -0.53] — Standard error of the least square mean
Statistical Analysis 20: Comparison: GFT505 120mg vs Placebo; Apo E/B; Test type: Superiority; p = 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.08, 95% CI 2-sided [-1.72 to -0.43] — Standard error of the least square mean

28. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Leptin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in leptin (to assess insulin resistance).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
ng/mL | -0.21 (9.55) | 3.51 (10.67) | 3.01 (8.08)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.066, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -2.8, 95% CI 2-sided [-5.79 to 0.18] — Least square mean changes from baseline
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.615, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.77, 95% CI 2-sided [-2.24 to 3.77] — Standard error of the least square mean

29. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Insulin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in insulin (to assess insulin resistance).
  Participants with missing data for Insulin at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 76
pmol/L | -33.88 (189.64) | -26.12 (111.76) | 8.92 (112.26)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.307, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -17.4, 95% CI 2-sided [-50.88 to 16.08] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.213, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -21.41, 95% CI 2-sided [-55.17 to 12.34] — Standard error of the least square mean

30. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: C Peptide
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in C peptide (to assess insulin resistance).
  Participants with missing data for C Peptide at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 77 | 76
nmol/L | -0.17 (0.55) | -0.03 (0.48) | 0.12 (0.58)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.23, 95% CI 2-sided [-0.37 to -0.08] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.068, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.14, 95% CI 2-sided [-0.29 to 0.01] — Standard error of the least square mean

31. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Homeostatic Model Assessment-insulin Resistance (HOMA-IR)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in homeostatic model assessment-insulin resistance (HOMA-IR; to assess insulin resistance).
  The HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (μU/ml) x fasting plasma glucose (mmol/l) / 22.5
  A decrease in HOMA-IR indicates a positive outcome. HOMA-IR values of greater than 1.9 indicates early insulin resistance and levels above 2.9 indicate significant insulin resistance.
  Participants with missing data for HOMA-IR at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 78 | 76
HOMA-IR score | -1.10 (10.76) | -1 (6.86) | 1.01 (4.96)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.448, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.8, 95% CI 2-sided [-2.86 to 1.27] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.267, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -1.17, 95% CI 2-sided [-3.25 to 0.9] — Standard error of the least square mean

32. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Free Fatty Acids (FFA)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in free fatty acids (FFA; to assess insulin resistance).
  Participants with missing data for Free Fatty Acids (FFA) at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 78 | 78 | 76
mmol/L | -0.04 (0.25) | -0.04 (0.24) | 0.05 (0.26)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.095, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.05, 95% CI 2-sided [-0.11 to 0.01] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.022, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.07, 95% CI 2-sided [-0.13 to -0.01] — Standard error of the least square mean

33. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Plasma Glucose
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in plasma glucose (to assess insulin resistance).
  Participants with missing data for Plasma Glucose at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 75
mmol/L | 0.17 (1.23) | 0.22 (1.70) | 0.67 (1.95)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.077, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.46, 95% CI 2-sided [-0.96 to 0.05] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.172, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.36, 95% CI 2-sided [-0.87 to 0.16] — Standard error of the least square mean

34. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Glycosylated Haemoglobin A1c (HbA1c)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in glycosylated haemoglobin A1c (HbA1c; to assess insulin resistance).
  Participants with missing data for Haemoglobin A1c (HbA1c) at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 81 | 77 | 77
percentage of HbA1c | 0.22 (0.56) | 0.03 (0.70) | 0.25 (0.69)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.732, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.04, 95% CI 2-sided [-0.24 to 0.17] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.062, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.2, 95% CI 2-sided [-0.4 to 0.01] — Standard error of the least square mean

35. Secondary Outcome: Changes From Baseline to Week 52 in Insulin Resistance: Fructosamine
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in Fructosamine (to assess insulin resistance).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
umol/L | 16.27 (27.53) | -8.24 (28.21) | 11.29 (28.62)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.4, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 3.66, 95% CI 2-sided [-4.89 to 12.2] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -16.22, 95% CI 2-sided [-24.99 to -7.44] — Standard error of the least square mean

36. Secondary Outcome: Changes From Baseline to Week 52 in Inflammatory Markers: Fibrinogen and Haptoglobin
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to Week 52, in fibrinogen and haptoglobin (inflammatory markers).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
g/L
  Fibrinogen: number analyzed (Participants) | 82 | 76 | 75
  Fibrinogen | -0.37 (0.70) | -0.37 (0.79) | -0.05 (0.66)
  Haptoglobin: number analyzed (Participants) | 81 | 77 | 76
  Haptoglobin | -0.19 (0.32) | -0.20 (0.40) | 0.09 (0.35)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Fibrinogen; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.36, 95% CI 2-sided [-0.54 to -0.17] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Fibrinogen; Test type: Superiority; p = 0.005, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.27, 95% CI 2-sided [-0.46 to -0.08]; Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Haptoglobin; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.25, 95% CI 2-sided [-0.35 to -0.15] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Haptoglobin; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.27, 95% CI 2-sided [-0.37 to -0.17] — Standard error of the least square mean

37. Secondary Outcome: Changes From Baseline to Week 52 in Inflammatory Markers: Tumour Necrosis Factor Alpha and Interleukine 6
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to Week 52, in tumour necrosis factor alpha and interleukine 6 (inflammatory markers).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
pg/mL
  Tumour Necrosis Factor alpha: number analyzed (Participants) | 81 | 78 | 77
  Tumour Necrosis Factor alpha | 1.37 (6.14) | -2.45 (38.58) | 0.19 (10.46)
  Interleukine 6: number analyzed (Participants) | 82 | 78 | 76
  Interleukine 6 | 0.37 (4.20) | -1.14 (10.33) | -0.06 (1.37)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Tumour Necrosis Factor alpha; Test type: Superiority; p = 0.742, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.57, 95% CI 2-sided [-2.9 to 4.06] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Tumour Necrosis Factor alpha; Test type: Superiority; p = 0.107, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 2.9, 95% CI 2-sided [-0.63 to 6.43] — Standard error of the least square mean
Statistical Analysis 3: Comparison: GFT505 80mg vs Placebo; Interleukine 6; Test type: Superiority; p = 0.362, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.5, 95% CI 2-sided [-0.58 to 1.59] — Standard error of the least square mean
Statistical Analysis 4: Comparison: GFT505 120mg vs Placebo; Interleukine 6; Test type: Superiority; p = 0.894, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.07, 95% CI 2-sided [-1.03 to 1.18] — Standard error of the least square mean

38. Secondary Outcome: Changes From Baseline to Week 52 in Inflammatory Markers: Plasminogen Activator Inhibitor 1 (PAI-1)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to Week 52, in plasminogen activator inhibitor 1 (PAI-1; inflammatory marker).
  Participants with missing data for Plasminogen Activator Inhibitor 1 (PAI-1) at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 68 | 77 | 66
ng/mL | -0.51 (3.51) | 0.21 (4.28) | -0.14 (4.74)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.229, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.76, 95% CI 2-sided [-2 to 0.48] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.463, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.45, 95% CI 2-sided [-1.67 to 0.76] — Standard error of the least square mean

39. Secondary Outcome: Changes From Baseline to Week 52 in Inflammatory Markers: C-Reactive Protein (CRP)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg or GFT505 120mg the changes from baseline to Week 52, in C-Reactive Protein (CRP; inflammatory marker).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set
Measure: Mean (Standard Deviation); unit: Log (mg/L)
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
Log (mg/L) | -0.04 (0.72) | -0.05 (0.81) | 0.20 (0.74)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.065, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.21, 95% CI 2-sided [-0.42 to 0.01] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.098, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.19, 95% CI 2-sided [-0.41 to 0.03] — Standard error of the least square mean

40. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Creatinine (Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in creatinine (safety markers; renal function parameter).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 89 | 92
μmol/L | 2.03 (7.89) | 5.61 (8.18) | 1.27 (7.85)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.553, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.7, 95% CI 2-sided [-1.61 to 3.01] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 4.31, 95% CI 2-sided [1.97 to 6.64] — Standard error of the least square mean

41. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Creatinine Clearance (Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in creatinine clearance (safety marker; renal function parameter).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 89 | 92
mL/min | -0.06 (0.94) | -0.56 (2.22) | -0.09 (0.62)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.861, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.04, 95% CI 2-sided [-0.37 to 0.44] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.052, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.4, 95% CI 2-sided [-0.81 to 0] — Standard error of the least square mean

42. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Uric Acid (Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in uric acid (safety marker; renal function parameter).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 89 | 92
mmol/L | 0 (0.06) | 0.01 (0.05) | -0.01 (0.06)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.473, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.01, 95% CI 2-sided [-0.01 to 0.02] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.124, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.01, 95% CI 2-sided [0 to 0.03] — Standard error of the least square mean

43. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Blood Urea Nitrogen (BUN; Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in blood urea nitrogen (BUN; safety marker; renal function parameter).
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol urea/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 89 | 92
mmol urea/L | 0.61 (1.28) | 0.67 (1.22) | -0.17 (1.14)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.81, 95% CI 2-sided [0.47 to 1.15] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.85, 95% CI 2-sided [0.5 to 1.19] — Standard error of the least square mean

44. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Cystatin C (Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in cystatin C (safety marker; renal function parameter).
  Participants with missing data for Cystatin C at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 87 | 89
mg/L | 0.05 (0.10) | 0.04 (0.22) | 0.04 (0.13)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.842, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0, 95% CI 2-sided [-0.04 to 0.04] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.589, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.01, 95% CI 2-sided [-0.03 to 0.05] — Standard error of the least square mean

45. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Beta2-microglobulin (Renal Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in beta2-microglobulin (safety marker; renal function parameter).
  Participants with missing data for Beta2-microglobulin at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 87 | 89
μg/L | -22.26 (326.42) | 0.11 (466.43) | -83.48 (279.31)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.325, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 48.93, 95% CI 2-sided [-8.73 to 146.6] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.066, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 93.21, 95% CI 2-sided [-6.06 to 192.49] — Standard error of the least square mean

46. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP; Cardiac Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in N-terminal prohormone of brain natriuretic peptide (NT-proBNP; safety marker; cardiac function parameter).
  Participants with missing data for NT-proBNP at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 93 | 87 | 89
pmol/L | 1.54 (4.16) | 0.38 (4.81) | -1.24 (5.35)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 2.41, 95% CI 2-sided [1.1 to 3.72] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 1.59, 95% CI 2-sided [0.26 to 2.91] — Standard error of the least square mean

47. Secondary Outcome: Changes From Baseline to Week 52 in Safety Markers: Troponin T (Cardiac Function Parameter)
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to week 52, in troponin T (safety marker; cardiac function parameter).
  Participants with missing data for Troponin T at baseline (Visit 2) or Visit 8 were not imputed in the analysis explaining the difference with the number of participants reported in the "Efficacy Evaluable Set" of the Participant Flow.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Safety population
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 92 | 87 | 89
μg/L | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.447, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0, 95% CI 2-sided [0 to 0] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.758, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0, 95% CI 2-sided [0 to 0] — Standard error of the least square mean

48. Secondary Outcome: Changes From Baseline to Week 52 in Body Weight
Description: To evaluate after 52 weeks of daily administration of GFT505 80mg, or GFT505 120mg, the changes from baseline to Week 52, in body weight.
Time Frame: Baseline (Visit 2; Week 0) to Visit 8 (Week 52)
Population: Efficacy evaluable set (EES)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
Number analyzed (Participants) | 82 | 78 | 77
kg | 0.11 (3.61) | -0.69 (4.09) | -0.04 (3.40)
Statistical Analysis 1: Comparison: GFT505 80mg vs Placebo; Test type: Superiority; p = 0.942, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = -0.04, 95% CI 2-sided [-1.12 to 1.04] — Standard error of the least square mean
Statistical Analysis 2: Comparison: GFT505 120mg vs Placebo; Test type: Superiority; p = 0.304, Mixed Models Analysis; Baseline parameter value and presence of diabetes as random factors; Difference in least square mean change = 0.57, 95% CI 2-sided [-0.52 to 1.66] — Standard error of the least square mean

ADVERSE EVENTS:
Time Frame: Adverse event information was collected at every study visit from screening up to the termination of the study corresponding to 64 weeks.
Description: The investigator established whether or not any adverse event had occurred at each visit (from the date of consent to the last study visit). The participant was questioned in a general manner to determine specific symptoms without offering the patient any suggestion. Serious adverse event reporting began from signature of the participant informed consent form and ended at the last study visit.
Arm/Group | GFT505 80mg | GFT505 120mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/89 | 0/92
Serious Adverse Events (participants affected / at risk) | 12/93 | 14/89 | 9/92
Other Adverse Events (participants affected / at risk) | 85/93 | 86/89 | 85/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GFT505 80mg (N=93) | GFT505 120mg (N=89) | Placebo (N=92)
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Device breakage (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Bladder diverticulum (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFT505 80mg (N=93) | GFT505 120mg (N=89) | Placebo (N=92)
Nausea (Gastrointestinal disorders) | 18 (23) | 17 (20) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 9 (11) | 13 (15)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 11 (12) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 9 (9) | 6 (6)
Vomiting (Gastrointestinal disorders) | 7 (8) | 8 (9) | 9 (12)
Constipation (Gastrointestinal disorders) | 7 (8) | 5 (5) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 2 (2) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Fatigue (General disorders) | 13 (15) | 12 (14) | 14 (16)
Chest pain (General disorders) | 4 (5) | 7 (7) | 3 (3)
Asthenia (General disorders) | 7 (10) | 0 (0) | 5 (6)
Influenza like illness (General disorders) | 1 (1) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 10 (11) | 6 (6) | 8 (8)
Nasopharyngitis (Infections and infestations) | 9 (13) | 5 (6) | 5 (5)
Influenza (Infections and infestations) | 10 (12) | 3 (3) | 5 (6)
Sinusitis (Infections and infestations) | 5 (5) | 9 (11) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (10) | 6 (6) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6) | 11 (11) | 10 (11)
Blood creatine phosphokinase increased (Investigations) | 4 (6) | 7 (7) | 2 (2)
Hepatic enzyme increased (Investigations) | 4 (4) | 3 (3) | 3 (3)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 4 (4) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 (7) | 4 (5) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 9 (9) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (10) | 6 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 6 (7)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (23) | 12 (14) | 15 (17)
Dizziness (Nervous system disorders) | 10 (12) | 6 (6) | 9 (9)
Anxiety (Psychiatric disorders) | 6 (7) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (5) | 1 (1)
Sleep disorder (Psychiatric disorders) | 5 (5) | 2 (2) | 4 (4)
Leukocyturia (Renal and urinary disorders) | 10 (12) | 8 (9) | 12 (17)
Glycosuria (Renal and urinary disorders) | 1 (1) | 6 (6) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 6 (6)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (5) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (8) | 6 (6) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 5 (5) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All materials, information (oral or written) and unpublished documentation provided to the Investigators (or any company/institution acting on their behalf) are the exclusive property of the Sponsor and may not be given or disclosed, either in part or in whole, by the Investigator or by any person under his/her authority to any third party without the prior express consent of the Sponsor.